CLINICAL TRIAL: NCT03673085
Title: A First in Human, Randomized, Double-blind, Single Ascending Dose, Phase Ia Clinical Study to Assess the Safety, Tolerability and Pharmacokinetic Parameters of CN128 Tablets in Thalassemia Patients Aged 16 and Above
Brief Title: Clinical Study of CN128 in Thalassemia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zede Pharma-Tech Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: D160605
Record Dates: First submitted 2018-03-15; First posted 2018-09-17 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Group 1-1 (Experimental): The dose of CN128 is 2.5 mg/kg bw.
  Interventions: Drug: CN128
- Group 1-2 (Placebo Comparator): The dose of placebo is 2.5 mg/kg bw.
  Interventions: Other: placebo
- Group 2-1 (Experimental): The dose of CN128 is 5 mg/kg bw.
  Interventions: Drug: CN128
- Group 2-2 (Placebo Comparator): The dose of placebo is 5 mg/kg bw.
  Interventions: Other: placebo
- Group 3-1 (Experimental): The dose of CN128 is 10 mg/kg bw.
  Interventions: Drug: CN128
- Group 3-2 (Placebo Comparator): The dose of placebo is 10 mg/kg bw.
  Interventions: Other: placebo
- Group 4-1 (Experimental): The dose of CN128 is 15 mg/kg bw.
  Interventions: Drug: CN128
- Group 4-2 (Placebo Comparator): The dose of placebo is 15 mg/kg bw.
  Interventions: Other: placebo
- Group 5-1 (Experimental): The dose of CN128 is 20 mg/kg bw.
  Interventions: Drug: CN128
- Group 5-2 (Placebo Comparator): The dose of placebo is 20 mg/kg bw.
  Interventions: Other: placebo
- Group 6-1 (Experimental): The dose of CN128 is 30 mg/kg bw.
  Interventions: Drug: CN128
- Group 6-2 (Placebo Comparator): The dose of placebo is 30 mg/kg bw.
  Interventions: Other: placebo
- Group 7-1 (Experimental): The dose of CN128 is 45 mg/kg bw.
  Interventions: Drug: CN128
- Group 7-2 (Placebo Comparator): The dose of placebo is 45 mg/kg bw.
  Interventions: Other: placebo
- Group 8-1 (Experimental): The dose of CN128 is 60 mg/kg bw.
  Interventions: Drug: CN128
- Group 8-2 (Placebo Comparator): The dose of placebo is 60 mg/kg bw.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: CN128 — CN128
  Arms: Group 1-1; Group 2-1; Group 3-1; Group 4-1; Group 5-1; Group 6-1; Group 7-1; Group 8-1
Other: placebo — The tablets without CN128
  Arms: Group 1-2; Group 2-2; Group 3-2; Group 4-2; Group 5-2; Group 6-2; Group 7-2; Group 8-2

SUMMARY:
1. Primary objectives:

   * To determine the maximum tolerated dose (MTD) of CN128 for single oral administration in thalassemia patients aged 16 and above
   * To study the pharmacokinetics of CN128 in thalassemia patients aged 16 and above
2. Design:

   The study is designed as a randomized, double-blind, single ascending dose, phase Ia (first in human) trial.

   The study is consisted of: single dose ascending; dose escalation pharmacokinetics; metabolite structure identification in plasma, urine and feces.
3. Subject inclusion criteria:

   * Thalassemia patients with serum ferritin ≥500 μg/L
   * Patients aged 16 and above
   * Without blood transfusion within 1 week before admission, with hemoglobin ≥ 80 g/L
   * Voluntarily participate in the experiment, and the process of obtaining informed consent form meeting the requirements of GCP
4. Subject exclusion criteria:

   * Hepatitis B surface antigen positive, hepatitis B core antibody positive and HBV-DNA positive, hepatitis C anti-HCV positive, HIV positive, Treponema pallidum positive
   * Patients with history of active digestive tract diseases (including gastric ulcer, duodenal ulcer, gastroesophageal varices, ulcerative colitis, Crohn's disease, digestive tract tumors, familial genetic multiple intestinal polyps), history of digestive tract perforation, history of digestive tract surgery and influence on drug absorption, and other patients whom investigators believe to have potential intestinal complications
   * Liver dysfunction (ALT or AST > 2.5×ULN); or renal dysfunction (serum creatinine > 1.5×ULN)
   * Uncontrolled active infections
   * Patients currently taking CYP3A strong inducer or inhibitor drugs or drugs that may prolong the QT interval without temporary suspension of use or temporary substitution of the said drugs
   * ect.
5. Usage:

   After fasting for at least 10 hours, the whole tablet was swallowed with 240 mL warm water on an empty stomach. Water was forbidden within 1 hour before and after the administration. Water was allowed 1 hour after administration.
6. Pharmacokinetic assessment of CN128 administration:

   PK parameters of CN128 include AUC 0-t, AUC 0-∞, Cmax, Tmax, t1/2, CL/F, Vd/F, MRT ,λz etc.
7. Safety and tolerability assessments:

   Evaluation was based on the incidence of adverse events (AE) after administration, termination information, laboratory test results, 12-lead electrocardiogram and vital signs.
8. Statistics

DETAILED DESCRIPTION:
1. Primary objectives:

   · To determine the maximum tolerated dose (MTD) of CN128 for single oral administration in thalassemia patients aged 16 and above

   · To study the pharmacokinetics of CN128 in thalassemia patients aged 16 and above
2. Design:

   The study is designed as a randomized, double-blind, single ascending dose, phase Ia (first in human) trial.

   The study is consisted of:

   · Single dose ascending: The trial will start with the lowest dose of CN128 given to 3 subjects, and the lowest dose of placebo given to 1 subjects (2.5 mg/kg body weight [bw], single dose).The dose of second group is 5 mg/kg bw.The dose of third group is 10 mg/kg bw.The dose of fourth group is 15 mg/kg bw.The dose of fifth group is 20 mg/kg bw.The dose of sixth group is 30 mg/kg bw.The dose of seventh group is 45 mg/kg bw.The dose of final group is 60 mg/kg bw.
   * Dose escalation pharmacokinetics:

   AUC 0-t, AUC 0-∞, Cmax, Tmax, t1/2, CL/F, Vd/F, MRT ,λz etc.

   · Metabolite structure identification in plasma, urine and feces: Collecting plasma, urine and feces samples for identifying CN128 metabolites in them.
3. Subject inclusion criteria:

   · Thalassemia patients with serum ferritin ≥500 μg/L
   * Patients aged 16 and above
   * Without blood transfusion within 1 week before admission, with hemoglobin ≥ 80 g/L
   * Voluntarily participate in the experiment, and the process of obtaining informed consent form meeting the requirements of GCP
4. Subject exclusion criteria:

   · Hepatitis B surface antigen positive, hepatitis B core antibody positive and HBV-DNA positive, hepatitis C anti-HCV positive, HIV positive, Treponema pallidum positive

   · Patients with history of active digestive tract diseases (including gastric ulcer, duodenal ulcer, gastroesophageal varices, ulcerative colitis, Crohn's disease, digestive tract tumors, familial genetic multiple intestinal polyps), history of digestive tract perforation, history of digestive tract surgery and influence on drug absorption, and other patients whom investigators believe to have potential intestinal complications

   · Liver dysfunction (ALT or AST > 2.5×ULN); or renal dysfunction (serum creatinine > 1.5×ULN)

   · Uncontrolled active infections

   · Patients currently taking CYP3A strong inducer or inhibitor drugs or drugs that may prolong the QT interval without temporary suspension of use or temporary substitution of the said drugs

   · Allergic constitution: allergic to or with contraindication of main ingredients or excipients of CN128 tablets (microcrystalline cellulose, cross-linked sodium carboxymethyl cellulose, silica, sodium stearate fumarate, Opadry)

   · Patients who have abnormal ECG with clinical significance: congenital long QT syndrome or known family history of long QT syndrome; QTc > 450ms (male) or QTc > 470ms (female); patients who have ventricular or atrial tachyarrhythmia with clinical significance, etc.

   · Family planning participants (including male subjects) during or within three months after the trial

   · Patients with a history of blood donation within 3 months before the trial

   · Patients with a history of smoking (more than 5 cigarettes or products with equivalent nicotine per day), alcoholism (more than 14 units of alcohol per week: 1 alcohol unit equals 10 mL or 8 g pure alcohol; 25 mL 40% liquor, 330 mL 5% beer, 175 mL 12% red wine equals 1.0, 1.5, 2.0 alcohol units respectively), drug abuse and addiction history

   · Patients who smoke, drink or eat any food containing alcohol, xanthine or grapefruit (including chocolate, tea, coffee or cola drinks) within 48 h before the using of test drug

   · The subject of any other clinical trials within 3 months before using of the test drug except for non interventional studies
   * Patients with positive results of nicotine and urine drug screening
   * Patients with difficult venous blood collection
   * Any patient with conditions which the investigators resume inappropriate to participate in this study, such as: poor health status, poor compliance, unwillingness or inability to comply with treatment regimens, including delayed visits
5. Usage:

   After fasting for at least 10 hours, the whole tablet was swallowed with 240 mL warm water on an empty stomach. Water was forbidden within 1 hour before and after the administration. Water was allowed 1 hour after administration.
6. Pharmacokinetic assessment of CN128 administration:

   PK parameters of CN128 include AUC 0-t, AUC 0-∞, Cmax, Tmax, t1/2, CL/F, Vd/F, MRT ,λz etc.
7. Safety and tolerability assessments:

   Evaluation was based on the incidence of adverse events (AE) after administration, termination information, laboratory test results, 12-lead electrocardiogram and vital signs.
8. Statistics:

   * Pharmacokinetic analysis:

Phoenix WinNonlin software (Pharsight Corporation, version 7.0) was used to estimate and analyze the parameters of PK in non-atrioventricular model according to dosage. The pharmacokinetic parameters were calculated in actual time to fully reflect the characteristics of drug absorption, distribution, metabolism and excretion in human body. The PK parameters of each participant were calculated according to the following methods. PK parameters include:

AUC0-t, AUC0-∞, Cmax, Tmax, t1/2, CL/F, Vd/F, MRT, λz; Descriptive statistics of untransformed data of drug concentration in plasma at each time point, AUC0 t, AUC0-∞, Cmax, Tmax, t1/2, CL/F, Vd/F, MRT and λz were summarized. Descriptive statistics was used in the analysis of Number (N), arithmetic mean, geometric mean, standard deviation (SD), CV, minimum, median and maximum.

· Linear correlation analysis for dosage: The dose dependence of Cmax, AUC0-t and AUC0-∞ was evaluated. Linear correlation analysis of main pharmacokinetic parameters and dosage was done for each subject by power model.

· Safety analysis: All AE, treatment emergent adverse events (TEAE), drug-related TEAE, grade 3 or above TEAE, serious adverse events (SAE), drug-related SAE, TEAE leading to death, TEAE leading to termination of trial, drug-relation TEAE leading to termination of trial and drug-related TEAE leading to discontinuation of use of test drug were summarized for case number, subject number and incidence rate. Summary of cases and incidence. P value for the incidence of these AEs with different classifications was calculated by Fisher's exact test.

TEAE, SAE, drug-related TEAE, drug-related SAE, TEAE leading to the termination of the trial, and TEAE leading to the discontinuation of drug use were summarized and described according to the system organ classification (SOC), preferred terminology (PT) and study group. The severity of TEAE and drug-related TEAE was also summarized according to SOC, PT and study groups.

The measured value of parameters and change of baseline of vital signs, 12-lead ECG, physical examination, clinical laboratory examination, etc. were summarized according to the planned time point and the study group.

Determine dose-limited toxicity of a single dose in human (DLT); Determine the maximum tolerated dose of a single dose in human (MTD).

ELIGIBILITY:
Subject inclusion criteria:

* Thalassemia patients with serum ferritin ≥500 μg/L
* Patients aged 16 and above
* Without blood transfusion within 1 week before admission, with hemoglobin ≥ 80 g/L
* Voluntarily participate in the experiment, and the process of obtaining informed consent form meeting the requirements of GCP

Subject exclusion criteria:

* Hepatitis B surface antigen positive, hepatitis B core antibody positive and HBV-DNA positive, hepatitis C anti-HCV positive, HIV positive, Treponema pallidum positive
* Patients with history of active digestive tract diseases (including gastric ulcer, duodenal ulcer, gastroesophageal varices, ulcerative colitis, Crohn's disease, digestive tract tumors, familial genetic multiple intestinal polyps), history of digestive tract perforation, history of digestive tract surgery and influence on drug absorption, and other patients whom investigators believe to have potential intestinal complications
* Liver dysfunction (ALT or AST > 2.5×ULN); or renal dysfunction (serum creatinine > 1.5×ULN)
* Uncontrolled active infections
* Patients currently taking CYP3A strong inducer or inhibitor drugs or drugs that may prolong the QT interval without temporary suspension of use or temporary substitution of the said drugs
* Allergic constitution: allergic to or with contraindication of main ingredients or excipients of CN128 tablets (microcrystalline cellulose, cross-linked sodium carboxymethyl cellulose, silica, sodium stearate fumarate, Opadry)
* Patients who have abnormal ECG with clinical significance: congenital long QT syndrome or known family history of long QT syndrome; QTc > 450ms (male) or QTc > 470ms (female); patients who have ventricular or atrial tachyarrhythmia with clinical significance, etc.
* Family planning participants (including male subjects) during or within three months after the trial
* Patients with a history of blood donation within 3 months before the trial
* Patients with a history of smoking (more than 5 cigarettes or products with equivalent nicotine per day), alcoholism (more than 14 units of alcohol per week: 1 alcohol unit equals 10 mL or 8 g pure alcohol; 25 mL 40% liquor, 330 mL 5% beer, 175 mL 12% red wine equals 1.0, 1.5, 2.0 alcohol units respectively), drug abuse and addiction history
* Patients who smoke, drink or eat any food containing alcohol, xanthine or grapefruit (including chocolate, tea, coffee or cola drinks) within 48 h before the using of test drug
* The subject of any other clinical trials within 3 months before using of the test drug except for non interventional studies
* Patients with positive results of nicotine and urine drug screening
* Patients with difficult venous blood collection
* Any patient with conditions which the investigators resume inappropriate to participate in this study, such as: poor health status, poor compliance, unwillingness or inability to comply with treatment regimens, including delayed visits

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Temperature | Day 1 to Day 8
  Vital signs checks
Change from baseline in Pulse | Day 1 to Day 8
  Vital signs checks; determine the patient's pulse which is one kind of physiological parameter
Change from baseline in Respiration | Day 1 to Day 8
  Vital signs checks; determine the patient's respiration which is one kind of physiological parameter
Change from baseline in Blood pressure | Day 1 to Day 8
  Vital signs checks; both systolic and diastolic will be measured
Skin examination | Day 1 to Day 8
  Physical examination
Change from baseline in Height | Day 1 to Day 8
  Physical examination
Change from baseline in Weight | Day 1 to Day 8
  Physical examination
Blood examination | Day 1 to Day 8
  Laboratory test: WBC, RBC, NEUT, BASO, etc.
Urine examination | Day 1 to Day 8
  Laboratory test: colour, appearance, glucose, protein, ketone, bilirubin, leukocyte, blood, and microscopic
Blood biochemical examination | Day 1 to Day 8
  Laboratory test: ALT, AST, ALP, LDH, AMS, BUN, ALB, etc.
Change from baseline in Serum iron | Day 1 to Day 8
  Laboratory test: Serum iron
Blood coagulation function | Day 1 to Day 8
  Laboratory test: fibrinogen, prothrombin time and corresponding INR, APTT
Electrocardiogram | Day 1 to Day 8
  Laboratory test: heart rate and QTc
Number of subjects with adverse events | Day 1 to Day 8
  Adverse events
AUC0-t of CN128 | 0h to 48h after study drug administration
  Pharmacokinetics parameters
AUC0-∞ of CN128 | 0h to 48h after study drug administration
  Pharmacokinetics parameters
Cmax of CN128 | 0h to 48h after study drug administration
  Pharmacokinetics parameters
t1/2 of CN128 | 0h to 48h after study drug administration
  Pharmacokinetics parameters
CL/F of CN128 | 0h to 48h after study drug administration
  Pharmacokinetics parameters
Vd/F of CN128 | 0h to 48h after study drug administration
  Pharmacokinetics parameters
MRT of CN128 | 0h to 48h after study drug administration
  Pharmacokinetics parameters: mean residence time

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Shentu, Principal Investigator — Single center
Locations (1):
- The first affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No